CLINICAL TRIAL: NCT02083926
Title: Ketamine Infusion for Social Anxiety Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patterson Trust Mentored Research Award: Clinical, Health Services and Policy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1310012947
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; SAD; Ketamine
MeSH Terms: conditions — Phobia, Social | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine infusion (Experimental): A ketamine infusion was given on day 0 (28) at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1 (1+28), 2 (2+28), 3 (3+28), 5 (5+28), 7 (7+28), 10 (10+28) and 14 (14+28) post-infusion.
  Interventions: Drug: Ketamine
- Saline infusion (Experimental): A saline infusion was given on day 0 (28) at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1 (1+28), 2 (2+28), 3 (3+28), 5 (5+28), 7 (7+28), 10 (10+28) and 14 (14+28) post-infusion.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ketamine — Ketamine (a single 0.5mg/kg intravenously over 40 minutes).
  Other Names: Ketalar
  Arms: Ketamine infusion
Other: Saline — Saline (a single 0.5mg/kg intravenously over 40 minutes).
  Other Names: Placebo
  Arms: Saline infusion

SUMMARY:
* Social Anxiety Disorder (SAD) is common and causes significant impairment.
* First-line treatments for Social Anxiety Disorder are only partially effective. Many SAD patients experience little or inadequate symptom relief with available treatments.
* Ketamine is a potent NMDA receptor antagonist. Ketamine represents an agent with a potentially novel mechanism of action for the treatment of anxiety disorders.
* Ketamine has demonstrated efficacy in the treatment of psychiatric disorders closely related to Social Anxiety Disorder including Major Depression, Bipolar Depression and possibly Obsessive-Compulsive Disorder.

Ketamine represents the possibility to provide rapid symptom relief to patients with SAD and may provide the mechanism for future drug development to treat SAD more rapidly and effectively.

DETAILED DESCRIPTION:
Roughly one-third to one-half of patients with generalized SAD do not experience significant clinical benefit from current evidence-based treatment for SAD such as pharmacotherapy with selective serotonin reuptake inhibitors (SSRI) or venlafaxine and cognitive behavioral therapy (CBT). Failure of anxiety relief in patients with SAD is a source of substantial morbidity, distress, and decreases in quality of life. Novel pharmacological treatments are needed to improve patient outcomes with SAD.

Converging lines of evidence from neuroimaging and pharmacological studies support the importance of glutamate abnormalities in the pathogenesis of SAD. In a Magnetic Resonance Spectroscopy (MRS) study, an elevated glutamate to creatinine ratio was found in the anterior cingulate cortex of SAD patients when compared to healthy controls. Elevated thalamic glutamine levels have been demonstrated in patients with SAD. Pre-clinical rodent studies have also established a strong link between glutamate regulation and anxiety.

Ketamine is a potent antagonist of the N-methyl-D-aspartate (NMDA) receptor, a major type of glutamate receptor in the brain. Ketamine is routinely used for anesthetic induction because of its dissociative properties. However in research studies, ketamine is effective treatment in reducing symptoms in depressive and possibly anxiety disorders. In multiple controlled clinical studies, ketamine has produced a rapid antidepressant effect in unipolar and bipolar depression. Ketamine's anti-depressant effects peak 1-3 days following infusion. Ketamine's antidepressant effect is observed long after ketamine has been metabolized and excreted by the body and after ketamine's sedative and dissociative effects have dissipated.

The results of several clinical studies suggest that ketamine may also have significant anxiolytic effects. Patients with major depressive disorder given a single ketamine infusion have shown strong and significant reductions in comorbid anxiety symptoms. A trial including 11 depressed patients demonstrated a significant reduction in anxiety symptoms (Hamilton Anxiety Rating Scale (HAM-A)) following ketamine infusion. This improvement is supported by one of the earlier placebo-controlled trials of ketamine which demonstrated that the psychic anxiety item was one of 4 (out of 21) items on the Hamilton Depression Rating Scale (HAM-D) demonstrating significant improvement after ketamine infusion.

The investigators goal is to conduct a randomized, placebo-controlled crossover study to explore the efficacy and time course of action of intravenous ketamine in the treatment of SAD.

ELIGIBILITY:
Inclusion Criteria:

1. Adult between the ages of 18 and 65 years
2. Meet DSM IV criteria for Social Anxiety Disorder by structured clinical interview (SCID) and have a LSAS >60 with or without co-morbid MDD

Exclusion Criteria:

1. Positive pregnancy test
2. History of substance abuse disorder within the last 6 months or positive urine toxicology on screening (within the previous 6 months).
3. History of pervasive developmental disorder or psychotic disorder by DSM-IV-TR criteria
4. Medical comorbidity that significantly increases the risks associated with ketamine infusion (e.g. untreated hypertension, significant cardiovascular disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdallah CG, Averill LA, Collins KA, Geha P, Schwartz J, Averill C, DeWilde KE, Wong E, Anticevic A, Tang CY, Iosifescu DV, Charney DS, Murrough JW. Ketamine Treatment and Global Brain Connectivity in Major Depression. Neuropsychopharmacology. 2017 May;42(6):1210-1219. doi: 10.1038/npp.2016.186. Epub 2016 Sep 8. PMID 27604566
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Davey HM, Barratt AL, Butow PN, Deeks JJ. A one-item question with a Likert or Visual Analog Scale adequately measured current anxiety. J Clin Epidemiol. 2007 Apr;60(4):356-60. doi: 10.1016/j.jclinepi.2006.07.015. Epub 2006 Dec 27. PMID 17346609
- [Background] Freitas-Ferrari MC, Hallak JE, Trzesniak C, Filho AS, Machado-de-Sousa JP, Chagas MH, Nardi AE, Crippa JA. Neuroimaging in social anxiety disorder: a systematic review of the literature. Prog Neuropsychopharmacol Biol Psychiatry. 2010 May 30;34(4):565-80. doi: 10.1016/j.pnpbp.2010.02.028. Epub 2010 Mar 4. PMID 20206659
- [Background] Glue P, Medlicott NJ, Harland S, Neehoff S, Anderson-Fahey B, Le Nedelec M, Gray A, McNaughton N. Ketamine's dose-related effects on anxiety symptoms in patients with treatment refractory anxiety disorders. J Psychopharmacol. 2017 Oct;31(10):1302-1305. doi: 10.1177/0269881117705089. Epub 2017 Apr 26. PMID 28441895
- [Derived] Taylor JH, Landeros-Weisenberger A, Coughlin C, Mulqueen J, Johnson JA, Gabriel D, Reed MO, Jakubovski E, Bloch MH. Ketamine for Social Anxiety Disorder: A Randomized, Placebo-Controlled Crossover Trial. Neuropsychopharmacology. 2018 Jan;43(2):325-333. doi: 10.1038/npp.2017.194. Epub 2017 Aug 29. PMID 28849779

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Infusion on Day 0, Saline Infusion on Day 28: A ketamine infusion was given on day 0 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1, 2, 3, 5, 7, 10 and 14 post-infusion. A saline infusion was given on Day 28 at a dose of 0.5mg/kg over a 40 minute period. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1+28, 2+28, 3+28, 5+28, 7+28, 10+28 and 14+28 post-infusion.
- Saline Infusion on Day 0, Ketamine Infusion on Day 28: A saline infusion was given on day 0 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1, 2, 3, 5, 7, 10 and 14 post-infusion. A Ketamine infusion was given on Day 28 at a dose of 0.5mg/kg over a 40 minute period. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1+28, 2+28, 3+28, 5+28, 7+28, 10+28 and 14+28 post-infusion.
Period: Overall Study
Arm/Group | Ketamine Infusion on Day 0, Saline Infusion on Day 28 | Saline Infusion on Day 0, Ketamine Infusion on Day 28
Started | 9 | 9
Completed | 8 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Infusion on Day 0, Saline Infusion on Day 28 | Saline Infusion on Day 0, Ketamine Infusion on Day 28 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.78 (13.50) | 28.67 (8.66) | 29.72 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 8 | 6 | 14
  Non-Hispanic Asian | 0 | 2 | 2
  Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Visual Analogue Scale for anxiety symptoms (VAS-anxiety) [Mean (Standard Deviation); unit: units on a scale] — Instrument that tries to measure anxiety, that is believed to range across a continuum of values and cannot easily be directly measured.We used a straight horizontal line of 100 mm in length. The ends were defined as the extreme limits of the parameter to be measured (anxiety); oriented from the left (no anxiety) to the right (worst anxiety ever felt). The patient marks on the line the point that they feel represents their perception of their current state.The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  units on a scale | 47.22 (18.89) | 57.78 (19.70) | 47.22 (18.89)
Liebowitz Social Anxiety Score (LSAS) [Mean (Standard Deviation); unit: units on a scale] — Clinician-administered scale for the assessment of fear and avoidance found in social phobia (SAD); it has 24 items divided into 2 subscales, 13 for performance anxiety, and 11 for social situations each rated from 0 to 3 (0=none,1=mild,2=moderate,3=definite). The sum scores for Fear and Avoidance results in an overall score (max 144 points). There are 4 clinician subscales: fear of social interaction, fear of performance, avoidance of social interaction and avoidance of performance 0 to 30= SAD is unlikely 30 to 60=SAD is probable 60 to 90=SADis very probable >90= SAD highly probable
  units on a scale | 93.89 (19.37) | 87.44 (14.53) | 90.67 (16.94)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale for Anxiety Symptoms (VAS-anxiety)
Description: Instrument that tries to measure anxiety, that is believed to range across a continuum of values and cannot easily be directly measured.We used a straight horizontal line of 100 mm in length. The ends were defined as the extreme limits of the parameter to be measured (anxiety); oriented from the left (no anxiety) to the right (worst anxiety ever felt). The patient marks on the line the point that they feel represents their perception of their current state.The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  We examined Visual Analog Scale (VAS) for anxiety symptoms at screening, 1 hour prior to infusion, 1, 2 and 3 hours after infusion, 1, 2, 3, 5, 7, 10, and 14 days following a single ketamine/saline infusion.
Time Frame: Day 1 (1+28)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketamine Infusion on Day 0 or Day 28: A ketamine infusion was given on day 0 or day 28 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1 (1+28), 2 (2+28), 3 (3+28), 5 (5+28), 7 (7+28), 10 (10+28) and 14 (14+28) post-infusion.
- Saline Infusion on Day 0 or Day 28: A saline infusion was given on day 0 or day 28 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, 1 (1+28), 2 (2+28), 3 (3+28), 5 (5+28), 7 (7+28), 10 (10+28) and 14 (14+28) post-infusion.
Arm/Group | Ketamine Infusion on Day 0 or Day 28 | Saline Infusion on Day 0 or Day 28
Number analyzed (Participants) | 18 | 17
units on a scale | 12.1 (18.6) | 19.6 (18.5)

2. Primary Outcome: Liebowitz Social Anxiety Score (LSAS)
Description: Clinician-administered scale for the assessment of fear and avoidance found in social phobia (SAD); it has 24 items divided into 2 subscales, 13 for performance anxiety, and 11 for social situations each rated from 0 to 3 (0=none,1=mild,2=moderate,3=definite). The sum scores for Fear and Avoidance results in an overall score (max 144 points). There are 4 clinician subscales: fear of social interaction, fear of performance, avoidance of social interaction and avoidance of performance 0 to 30= SAD is unlikely 30 to 60=SAD is probable 60 to 90=SADis very probable >90= SAD highly probable
Time Frame: Day 1 (1+28)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Saline Infusion on Day 0 or Day 28: A saline infusion was given on day 0 or day 28 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1 (1+28), 2 (2+28), 3 (3+28), 5 (5+28), 7 (7+28), 10 (10+28) and 14 (14+28) post-infusion.
Arm/Group | Ketamine Infusion on Day 0 or Day 28 | Saline Infusion on Day 0 or Day 28
Number analyzed (Participants) | 18 | 17
score on a scale | 66.1 (30.9) | 86.1 (30)

ADVERSE EVENTS:
Time Frame: 1 hour after infusion
Description: The Clinician-Administered Dissociative State Scale (CADSS) is a 27-item scale. The subjective component consists of 19 clinician administered items that are meant to depict the subjects state at the time that the items are being asked of them. The range of possible responses: 0 = not at all, 1 = slightly, 2= moderately, 3 = considerably, 4 = extremely. The clinician rates the 8 subjective items.
Groups:
- Ketamine Infusion on Day 0 or Day 28: Participants were randomized to receive ketamine either on day 0 or on day 28. The ketamine infusion was given at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1, 2, 3, 5, 7, 10 and 14 post-infusion.
- Saline Infusion on Day 0 or Day 28: Participants were randomized to receive a saline infusion either on day 0 or on day 28 at a dose of 0.5mg/kg over 40 minutes. Assessments were conducted pre-infusion, 3-h post-infusion, and days 1, 2, 3, 5, 7, 10 and 14 post-infusion.
Arm/Group | Ketamine Infusion on Day 0 or Day 28 | Saline Infusion on Day 0 or Day 28
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 15/18 | 4/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Infusion on Day 0 or Day 28 (N=18) | Saline Infusion on Day 0 or Day 28 (N=17)
things seem to be moving (Nervous system disorders) | 7 (7) | 2 (2)
things seem unreal (Nervous system disorders) | 9 (9) | 3 (3)
feel like you are separated from reality (Nervous system disorders) | 3 (3) | 1 (1)
looking at things outside of your body (Nervous system disorders) | 4 (4) | 0 (0)
Feel like a spectator (Nervous system disorders) | 7 (7) | 2 (2)
Feel disconnected from your own body (Nervous system disorders) | 5 (5) | 2 (2)
Sense of your own body feel changed (Nervous system disorders) | 4 (4) | 0 (0)
Objects look different (Nervous system disorders) | 3 (3) | 0 (0)
Feel as if you were in a tunnel (Nervous system disorders) | 5 (5) | 1 (1)
Things happening very quickly (Nervous system disorders) | 1 (1) | 1 (1)
Things you can't account for (Nervous system disorders) | 6 (6) | 1 (1)
Spaced out (Nervous system disorders) | 13 (13) | 4 (4)
Sounds almost disappear (Nervous system disorders) | 5 (5) | 1 (1)
things seem to be very real (Nervous system disorders) | 3 (3) | 0 (0)
Outside of your body (Nervous system disorders) | 4 (4) | 1 (1)
Colors seem brighter (Nervous system disorders) | 1 (1) | 1 (1)
Confused about who you really are (Nervous system disorders) | 2 (2) | 0 (0)
Parts of your body that don't fit together (Nervous system disorders) | 1 (1) | 0 (0)
gaps in your memory (Nervous system disorders) | 8 (8) | 0 (0)
having more than one identity (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0) — >100 beats per minute
diastolyc hypertension (Cardiac disorders) | 3 (3) | 0 (0) — >90 mm Hg (max of 106mm Hg)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
systolic hypertension (Cardiac disorders) | 2 (2) | 0 (0) — >160 mm Hg (max of 184mm Hg)
diastolyc hypotension (Cardiac disorders) | 2 (2) | 0 (0) — <60 mm Hg (min 49 mm Hg)
parestesias and numbness (Nervous system disorders) | 9 (9) | 0 (0)
dizziness (Nervous system disorders) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
A significant limitation of our study was that 17 of 18 subjects correctly identified when they received ketamine, suggesting that the use of saline as a placebo control for ketamine led to inadequate blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02083926/Prot_SAP_000.pdf